CLINICAL TRIAL: NCT02215681
Title: Acupuncture Effect on Inflammatory Markers in Pediatric Otitis Media With Effusion: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-13-ziv
Record Dates: First submitted 2014-07-09; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Otitis Media With Effusion
Keywords: otitis media with effusion; acupuncture; inflammatory markers
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): acupuncture treatment
  Interventions: Device: acupuncture
- standard treament (No Intervention): watchful waiting

INTERVENTIONS:
Device: acupuncture
  Arms: acupuncture

SUMMARY:
Objective: to evaluate acupunctures effect on inflammatory markers in pediatric Otitis Media with Effusion Methods: 100 Children with otitis media with effusion (OME) diagnosis, who are in watchful waiting for 3 month, will be randomized in two groups: acupuncture and control. 50 Children in the acupuncture group will receive standard treatment combined with acupuncture for 3 months. 50 Children in the control group will receive standard treatment only, for the same time period. After 3 months, both groups will be reassessed for OME. Children with no improvement from both groups will be assigned for tympanostomy.

Data collection: in children undergoing tympanostomy, middle ear effusion (MEE) will be collected, analyzed and evaluated for group differences.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy children ages 2-8 years
* autoscopic OME diagnosis
* tympanometry type B
* conductive hearing impairment of 30 decibel or more
* who are at watchful waiting treatment for 3 months
* signed parental consent.

Exclusion Criteria:

* lack of parental consent
* known coagulopathy
* past tympanostomy
* regular intake of steroids or cytotoxic drugs

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
presence of inflammatory markers in middle ear effusion | 3 months
  after 3 months, patients in both groups will be reevaluated for OME by micro otoscopy and tympanometry, including an audiogram. patients with no improvement, will be submitted for tympanostomy in accordance with standard criteria. middle ear effusion will be collected and analysed by ELISA for viral/bacterial RNA presence and flow cytometry for leukocyte presence. results will be statistically processed for between group differences.

SECONDARY OUTCOMES:
acupuncture effect on OME | 3 months
  after 3 months, patients from both group will undergo micro otoscopy,tympanometry and an audiogram to evaluate OME presence. group differences will be statistically processed

OTHER OUTCOMES:
acupuncture acceptance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: peter Gilbey, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel